CLINICAL TRIAL: NCT05371145
Title: Carnosine for Peripheral Arterial Disease Patients (Car-PAD)
Brief Title: Carnosine for Peripheral Arterial Disease Patients
Acronym: CAR-PAD
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shahid Baba (Other)
Responsible Party: Sponsor-Investigator, Shahid Baba, Assistant Professor, University of Louisville
Organization: University of Louisville (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 22.0098
Record Dates: First submitted 2022-04-29; First posted 2022-05-12 (Actual); Last update posted 2024-07-22 (Actual); Status verified 2024-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease | interventions — Carnosine

STUDY DESIGN:
Intervention Model Description: In a single arm open labelled safety trial, we will supplement carnosine for 3 months to subjects with non-claudication and claudication peripheral arterial disease (PAD), and determine if it improves walking ability. In our pilot study, we will enroll 20 male subjects measure the distance covered on the 6-minute walk test and the pain free walking capacity on the treadmill before, at baseline, and three months after carnosine supplementation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carnosine intervention for patients with PAD (Experimental): This is a single arm open labelled safety trial, where we will supplement carnosine for 3 months to subjects with non-claudication and claudication peripheral arterial disease (PAD), and determine if it improves walking ability.
  Interventions: Biological: Carnosine

INTERVENTIONS:
Biological: Carnosine — Determine whether carnosine supplementation (2 g/day) for 3 months in peripheral arterial disease patients improves 6MWT ability.

SUMMARY:
Oral supplementation of L-carnosine will increase muscle carnosine, stabilize HIF1-alpha promote angiogenesis, and thus improve the functioning of lower extremities in PAD patients.

DETAILED DESCRIPTION:
Peripheral arterial disease (PAD) is caused by atherosclerotic occlusion of the lower extremities that reduces blood flow and leads to intermittent claudication and critical limb ischemia. PAD is diagnosed by calculating the ratio of blood pressure at the ankle to that of the arm (the ankle-brachial index [ABI]). An ABI of <0.90 is indicative of atherosclerosis in the leg. Recent data from developed and developing countries have estimated that >200 million people worldwide and approximately 12 million people in United States have PAD3. Both symptomatic and asymptomatic PAD patients have an increased risk of mortality, morbidity, and a lower quality of life. With the increasing incidence of type 2 diabetes (T2D) and a rising aging population, the number of PAD patients is likely to increase. Because PAD is an under-recognized disease, currently few medications are available to improve the functional performance of these patients. Although surgical revascularization is an available treatment, grafts can fail and the stenosis can reoccur in these patients. To adequately compensate the loss of tissue due to occlusion, the current emphasis is to increase the therapeutic angiogenesis and arteriogenesis in the ischemic limb that could improve the walking ability and the quality of life in PAD patients. In a recent pre-clinical study it was shown that supplementation of carnosine(β-alanine-histidine) (500 mg/day) in heart failure patients for 6 months improves their performance on the 6-minute walking test (6MWT) compared with placebo-treated patients. Carnosine is a histidyl dipeptide present in high concentration in the skeletal muscle, brain, and heart. It is a food constituent that is present in red meat, chicken, and turkey. This dipeptide is synthesized by the ATP grasp enzyme carnosine synthetase and hydrolyzed to β-alanine and histidine by the serum and kidney carnosinase. Carnosine has the abilities to quench reactive aldehydes, bind metals, and buffer intracellular pH7. Numerous studies have shown that the supplementation of beta-alanine or carnosine increases the levels of carnosine in the skeletal muscle and improves the exercise performance in humans. Our preliminary studies with the mice model of hind limb ischemia (HLI) showed that both the pretreatment and supplementation of carnosine after femoral artery ligation increased blood flow in the ischemic limb compared with the non-treated mice. Mechanistic studies showed that the metal quenching ability of carnosine increased the expression of angiogenic factor VEGF and endothelial progenitor cells mobilization in the carnosine treated HLI mice. Similarly, the stabilization of HIF-1α, the master regulator of angiogenesis and angiogenic factor VEGF, was increased in the hypoxic C2C12 cells (murine myoblasts). Based on these pre-clinical studies, in this study PAD subjects will be recruited and supplemented with carnosine (2 g/day) for 3 months to examine if its supplementation improves walking performance compared with the baseline. Further, we will examine whether the supplementation of carnosine increases the capacity of pain-free treadmill walking time, extrusion of oxidative stress markers and mobilizes the endothelial progenitor cells in the blood.

ELIGIBILITY:
Inclusion Criteria:

1. Male subjects more than >50 to <80 years of age.
2. White or African American race.
3. English Speaking.
4. ABI 0.4-< 0.60
5. Willing to comply with protocol requirements.
6. Able to provide informed consent. -

Exclusion Criteria:

1. Subjects with HIV, hepatitis, significant liver disease, active infection, anemia, organ transplant, renal disease requiring dialysis, lung disease requiring oxygen, significant congenital heart disease, cancer of any type, and untreated thyroid disease.
2. Diagnosis of carnosinemia.
3. Known allergy to L-carnosine or meat.
4. Presence of a pacemaker.
5. Obesity from a known genetic defect.
6. Dementia.
7. Critical limb ischemia with below or above knee amputations.
8. Foot ulcers.
9. Major amputations.
10. Participating in other clinical trials.
11. End stage renal disease.
12. Presence of significant injury within 30 days before enrollment.
13. Prisoners.
14. Any metallic implants.
15. Poorly controlled diabetes (HbA1C >9%) -

Ages: 50 Years to 80 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2024-12-30 (Estimated)

PRIMARY OUTCOMES:
Carnosine for Peripheral Arterial Disease patients | One year
  Compare the effects of carnosine supplementation on the 6-minute walk test (6MWT) at the baseline and after three months of carnosine supplementation.
  Measure the total walking distance and compare the walking distance covered by the subjects at the start and completion of carnosine supplementation

SECONDARY OUTCOMES:
Graded treadmill test | one year
  Measure the onset of claudication onset time and peak walk time

CONTACTS AND LOCATIONS:
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Annex BH. Therapeutic angiogenesis for critical limb ischaemia. Nat Rev Cardiol. 2013 Jul;10(7):387-96. doi: 10.1038/nrcardio.2013.70. Epub 2013 May 14. PMID 23670612
- [Result] Hiatt WR, Hoag S, Hamman RF. Effect of diagnostic criteria on the prevalence of peripheral arterial disease. The San Luis Valley Diabetes Study. Circulation. 1995 Mar 1;91(5):1472-9. doi: 10.1161/01.cir.91.5.1472. PMID 7867189
- [Result] Criqui MH, Aboyans V. Epidemiology of peripheral artery disease. Circ Res. 2015 Apr 24;116(9):1509-26. doi: 10.1161/CIRCRESAHA.116.303849. PMID 25908725
- [Result] Lombardi C, Carubelli V, Lazzarini V, Vizzardi E, Bordonali T, Ciccarese C, Castrini AI, Dei Cas A, Nodari S, Metra M. Effects of oral administration of orodispersible levo-carnosine on quality of life and exercise performance in patients with chronic heart failure. Nutrition. 2015 Jan;31(1):72-8. doi: 10.1016/j.nut.2014.04.021. Epub 2014 May 10. PMID 25287762
- [Result] Drozak J, Veiga-da-Cunha M, Vertommen D, Stroobant V, Van Schaftingen E. Molecular identification of carnosine synthase as ATP-grasp domain-containing protein 1 (ATPGD1). J Biol Chem. 2010 Mar 26;285(13):9346-9356. doi: 10.1074/jbc.M109.095505. Epub 2010 Jan 22. PMID 20097752
- [Result] Teufel M, Saudek V, Ledig JP, Bernhardt A, Boularand S, Carreau A, Cairns NJ, Carter C, Cowley DJ, Duverger D, Ganzhorn AJ, Guenet C, Heintzelmann B, Laucher V, Sauvage C, Smirnova T. Sequence identification and characterization of human carnosinase and a closely related non-specific dipeptidase. J Biol Chem. 2003 Feb 21;278(8):6521-31. doi: 10.1074/jbc.M209764200. Epub 2002 Dec 6. PMID 12473676
- [Result] Hipkiss AR. Energy metabolism, proteotoxic stress and age-related dysfunction - protection by carnosine. Mol Aspects Med. 2011 Aug;32(4-6):267-78. doi: 10.1016/j.mam.2011.10.004. Epub 2011 Oct 15. PMID 22020113
- [Result] Harris RC, Stellingwerff T. Effect of beta-alanine supplementation on high-intensity exercise performance. Nestle Nutr Inst Workshop Ser. 2013;76:61-71. doi: 10.1159/000350258. Epub 2013 Jul 25. PMID 23899755
- [Result] Caruso J, Charles J, Unruh K, Giebel R, Learmonth L, Potter W. Ergogenic effects of beta-alanine and carnosine: proposed future research to quantify their efficacy. Nutrients. 2012 Jul;4(7):585-601. doi: 10.3390/nu4070585. Epub 2012 Jun 26. PMID 22852051
- [Result] Roger VL, Go AS, Lloyd-Jones DM, Adams RJ, Berry JD, Brown TM, Carnethon MR, Dai S, de Simone G, Ford ES, Fox CS, Fullerton HJ, Gillespie C, Greenlund KJ, Hailpern SM, Heit JA, Ho PM, Howard VJ, Kissela BM, Kittner SJ, Lackland DT, Lichtman JH, Lisabeth LD, Makuc DM, Marcus GM, Marelli A, Matchar DB, McDermott MM, Meigs JB, Moy CS, Mozaffarian D, Mussolino ME, Nichol G, Paynter NP, Rosamond WD, Sorlie PD, Stafford RS, Turan TN, Turner MB, Wong ND, Wylie-Rosett J; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart disease and stroke statistics--2011 update: a report from the American Heart Association. Circulation. 2011 Feb 1;123(4):e18-e209. doi: 10.1161/CIR.0b013e3182009701. Epub 2010 Dec 15. PMID 21160056